CLINICAL TRIAL: NCT05905731
Title: Study Evaluating the Safety and Efficacy of Autologous T-cells Transfected With mRNA Encoding Hepatitis-B Virus (HBV)-Antigen-specific T Cell Receptor (TCR) in Combination With Nucleos(t)Ide Analogue (NUC) for Chronic Hepatitis B
Brief Title: Autologous T-cells Transfected With mRNA Encoding HBV-TCR T Cell Therapy in Combination With NUC for Chronic Hepatitis B
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTCR-CHB-2-1
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HBV-TCR T cell infusion (Experimental): Autologous HBV specific TCR redirected T cells
  Interventions: Biological: TCR-T

INTERVENTIONS:
Biological: TCR-T — Stage-1: Patients will receive three biweekly HBV-TCR T cell infusions at escalating doses, ranging from 1 x 10^5 cells/kg to 5 x 10^6 cells/kg bodyweight (by IV infusion). Patients are to remain on existing HBV NUC treatment.
  Stage-2: Patients will receive three biweekly HBV-TCR T cell infusions at maximum dose as determined in Stage-1 study. Patients are to remain on existing HBV NUC treatment.

SUMMARY:
This is a single center, single arm, open label study to assess the safety, tolerability and effectiveness of the autologous HBV specific T cell receptor (HBV-TCR) redirected T cells in patients with chronic hepatitis B with ongoing with nucleos(t)ide analogue (NUC) treatment. This study will be conducted sequentially starting with Stage-1, followed by Stage-2.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg Positive, HBeAg Negative, Anti-HBe Positive (with HBeAg seroconversion).
* On first-line treatment with oral nucleoside analogs antiviral drug therapy for more than a year.
* Adequate organ function
* Willing to stop and/or not to be on other immunomodulators during the study period, and to inform in time when other treatments such as glucocorticoids are needed
* Liver biopsy, Fibroscan® or equivalent test obtained within the past 6 months demonstrating liver disease consistent with chronic HBV infection without evidence of bridging fibrosis or cirrhosis (≥ Metavir 3, recommended cut-off for Fibroscan 9.0kPa)
* Females of childbearing potential must have a negative pregnancy test at Screening (within 3 days prior to first dose) and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy. Willing and able to comply with all study procedures.
* Willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures.

Exclusion Criteria:

* History of Acute infection, gastrointestinal bleeding, etc. occurring within 28 days prior to study enrollment.
* Advanced liver cirrhosis, Child-Pugh score ≥ 7 or clinical symptoms of liver function decompensation such as ascites and varicose veins
* Positive test for other viral infections, anti-HAV IgM, anti HCV, anti-HDV, anti -HEV and anti-HIV Any item is positive; liver disease caused by other reasons (such as autoimmune liver disease, alcoholic liver disease, non-alcoholic liver disease, drug-induced liver disease and other liver diseases of unknown cause, etc.).
* History of or suspicion of hepatocellular carcinoma or alpha fetoprotein (AFP) > 20 ng/mL at Screening. If AFP > 20 ng/mL, hepatic imaging must exclude hepatocellular carcinoma.
* History of having received (in the last 6 months) or currently receiving any other cell therapies
* History of organ transplantation
* History of severe allergic reaction (hives or anaphylaxis) to blood products
* History of any Grade 4 immune-related AE from prior immunotherapy. Any immune-related AE that led to permanent discontinuation that occurred less than 6 months prior to leukapheresis or whole blood collection for production
* Use of any investigational product (IP) within 28 days of study treatment administration.
* Lack of peripheral venous or central venous access or any condition that would interfere with drug administration or collection of study samples

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation of HBV-TCR T cell treatment | Start of Treatment until 28 days post last dose
  Incidence of adverse events/serious adverse events

SECONDARY OUTCOMES:
To evaluate the capability of HBV-TCR T cell treatment to lower the levels of serum HBsAg | Start of treatment until 12 months post treatment follow-up
  This is based on quantitative changes of HBsAg levels from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, MD, Principal Investigator — Beijing 302 Hospital
Locations (1):
- The Fifth Medical Center of PLA General Hospital, Beijing, China